CLINICAL TRIAL: NCT00068445
Title: The Efficacy of Lamotrigine in the Management of Chemotherapy-Induced Peripheral Neuropathy: A Phase III Randomized, Double Blind, Placebo-Controlled Trial
Brief Title: Lamotrigine in Treating Peripheral Neuropathy Caused by Chemotherapy in Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N01C3; CDR0000322830 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Neurotoxicity; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: neurotoxicity; pain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neurotoxicity Syndromes; Pain | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I - lamotrigine (Experimental): Patients receive oral lamotrigine once daily for 2 weeks and then twice daily for 8 weeks. Treatment continues for 10 weeks in the absence of unacceptable toxicity.
  Quality of life, pain, mood states, and symptom distress are assessed at baseline and at 4, 6, 8, and 10 weeks.
  Patients are followed at 3-7 days.
  Interventions: Drug: lamotrigine
- Arm II - placebo (Other): Patients receive oral placebo once daily for 2 weeks and then twice daily for 8 weeks.
  Treatment continues for 10 weeks in the absence of unacceptable toxicity.
  Quality of life, pain, mood states, and symptom distress are assessed at baseline and at 4, 6, 8, and 10 weeks.
  Patients are followed at 3-7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: lamotrigine
  Arms: Arm I - lamotrigine
Other: Placebo
  Arms: Arm II - placebo

SUMMARY:
RATIONALE: Lamotrigine may be effective in reducing pain, numbness, tingling, and other symptoms of peripheral neuropathy. It is not yet known whether lamotrigine is effective in treating peripheral neuropathy caused by chemotherapy.

PURPOSE: This randomized phase III trial is studying how well lamotrigine works in reducing pain, numbness, tingling, and other symptoms of peripheral neuropathy caused by chemotherapy in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of lamotrigine vs placebo in reducing pain and symptoms of chemotherapy-induced peripheral neuropathy in patients with cancer.
* Compare symptom distress, mood states, functional abilities, and overall quality of life of patients treated with these agents.
* Determine the toxic effects of lamotrigine in these patients.

OUTLINE: This is a randomized, placebo-controlled, double-blind study. Patients are stratified according to neurotoxic chemotherapy received (taxanes vs platinum-based compounds vs vinca alkaloids vs combination vs other), status of neurotoxic chemotherapy (actively receiving therapy vs discontinued or completed), and duration of pain or neuropathy symptoms (1-3 months vs 3-6 months vs more than 6 months). Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Received, or are currently receiving, neurotoxic chemotherapy, including any of the following:

  * Taxanes (e.g., paclitaxel or docetaxel)
  * Platinum-based compounds (e.g., carboplatin, cisplatin, or oxaliplatin)
  * Vinca alkaloids (e.g., vincristine or vinblastine)
* Experiencing pain or symptoms of peripheral neuropathy for at least 1 month attributed to chemotherapy

  * Average daily pain rating of at least 4 out of 10 OR
  * Peripheral neuropathy at least grade 1 out of 3 using ECOG sensory neuropathy rating

PATIENT CHARACTERISTICS:

Age

* 18 and over

Life expectancy

* At least 6 months

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction or intolerance to lamotrigine
* No extreme difficulty swallowing pills
* No other identified causes of painful paresthesia preceding chemotherapy, including any of the following:

  * Radiation or malignant plexopathy
  * Lumbar or cervical radiculopathy
  * Pre-existing peripheral neuropathy of another etiology, such as any of the following:

    * Cyanocobalamin deficiency
    * AIDS
    * Monoclonal gammopathy
    * Diabetes
    * Heavy metal poisoning amyloidosis
    * Syphilis
    * Hyperthyroidism or hypothyroidism
    * Inherited neuropathy
* No significant psychiatric illness (e.g., mania, psychosis, or schizophrenia) that would preclude study participation
* Able to complete questionnaires

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics
* More than 7 days since prior methotrexate or other dihydrofolate inhibitors

Other

* More than 7 days since prior, and no concurrent use of any of the following:

  * Tricyclic antidepressants (e.g., amitriptyline, nortriptyline, or desipramine)

    * Concurrent selective serotonin reuptake inhibitors allowed
  * Monoamine oxidase inhibitors
  * Opioid analgesics
  * Anticonvulsants (e.g., gabapentin, topiramate, valproic acid, or clonazepam)
  * Adjuvant analgesics (e.g., mexiletine)

    * Prior nonsteroidal anti-inflammatory drugs allowed
  * Topical analgesics (e.g., lidocaine gel or patch) to the affected area
  * Amifostine
* More than 30 days since prior investigational agents for pain control
* No other concurrent investigational agents for pain control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2004-02; Primary Completion 2006-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi D. Rao, MD, MBBS, Study Chair — Mayo Clinic
Locations (23):
- United States (23):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates at June E. Nylen Cancer Center, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin

REFERENCES:
- [Result] Rao RD, Flynn PJ, Sloan JA, Wong GY, Novotny P, Johnson DB, Gross HM, Renno SI, Nashawaty M, Loprinzi CL. Efficacy of lamotrigine in the management of chemotherapy-induced peripheral neuropathy: a phase 3 randomized, double-blind, placebo-controlled trial, N01C3. Cancer. 2008 Jun 15;112(12):2802-8. doi: 10.1002/cncr.23482. PMID 18428211

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I - Lamotrigine: Patients receive oral lamotrigine (25 mg per pill) once daily for 2 weeks and then twice daily for 8 weeks. Treatment continues for 10 weeks total in the absence of unacceptable toxicity.
- Arm II - Placebo: Patients receive oral placebo once daily for 2 weeks and then twice daily for 8 weeks. Treatment continues for 10 weeks total in the absence of unacceptable toxicity.
Period: Randomization
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Started | 65 | 66
Completed | 63 | 62
Not Completed | 2 | 4
Not completed — Cancel | 1 | 3
Not completed — Ineligible | 1 | 1
Period: Treatment
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Started | 63 | 62
Completed | 34 | 46
Not Completed | 29 | 16
Not completed — Refused Further Treatment | 13 | 10
Not completed — Adverse Event | 7 | 1
Not completed — Other (Specifics not available) | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo | Total
Number analyzed (Participants) | 63 | 62 | 125
Age, Continuous [Mean (Full Range); unit: years] | 62 [29 to 84] | 59 [34 to 82] | 61 [29 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 27 | 24 | 51
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 62 | 125

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daily Pain Score as Measured Using a Pain Intensity Rating (NRS)
Description: The change in mean score for average daily pain from baseline to week 10 using the Pain Intensity Rating (NRS) are reported below. The NRS scale ranges from 0 to 10 with higher scores corresponding to having more pain.
Time Frame: From baseline to week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Number analyzed (Participants) | 34 | 46
units on a scale | -0.3 (2.76) | -0.5 (2.34)
Statistical Analysis 1: Comparison: Arm I - Lamotrigine vs Arm II - Placebo; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Average Pain Score as Measured Using the European Cooperative Oncology Group (ECOG) Neuropathy Scale (ENS)
Description: The change in mean score for average daily pain from baseline to week 10 using the European Cooperative Oncology Group (ECOG) neuropathy scale (ENS) are reported below. The ENS scale goes from 0 to 3 with 0=none, 1=mild paresthesias, 2=mild or moderate sensory loss and/or moderate paresthesias, and 3=severe sensory loss or paresthesias that interfere with function.
Time Frame: From baseline to week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Number analyzed (Participants) | 34 | 46
units on a scale | -0.4 (0.73) | -0.3 (1.00)
Statistical Analysis 1: Comparison: Arm I - Lamotrigine vs Arm II - Placebo; Test type: Superiority; p = 0.36, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: The Change in Overall Quality of Life as Measured by the Uniscale QOL From Baseline to Week 10
Description: The change in overall quality of life as measured by the Uniscale QOL (Week 10 minus Baseline) using the Wilcoxon test is reported for each arm below. The Uniscale is a score that ranges from 0 to 100, with 0 being QOL as bad as it can be and 100 being as good as it can be.
Time Frame: From baseline to week 10
Population: Participants with Uniscale QOL data at both time points available were assessed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Number analyzed (Participants) | 30 | 34
units on a scale | -4.3 (25.15) | 0.3 (22.09)
Statistical Analysis 1: Comparison: Arm I - Lamotrigine vs Arm II - Placebo; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Brief Pain Inventory (BPI) Worst Pain Score [Week 10 Minus Baseline]
Description: The average change in Brief Pain Inventory (BPI) Worst Pain scores between baseline and week 10 using Wilcoxon test are reported for each arm below. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: From baseline to week 10
Population: Participants with BPI Worst Pain data at both time points available were assessed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Number analyzed (Participants) | 27 | 36
units on a scale | 0.1 (3.17) | -0.6 (2.31)
Statistical Analysis 1: Comparison: Arm I - Lamotrigine vs Arm II - Placebo; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Brief Pain Inventory (BPI) Least Pain Score [Week 10 Minus Baseline]
Description: The average change in Brief Pain Inventory (BPI) Least Pain scores between baseline and week 10 using Wilcoxon test are reported for each arm below. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
  Time Frame:
  Up to 1 week post-treatment
Time Frame: From baseline to week 10
Population: Participants with BPI Least Pain data at both time points available were assessed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Number analyzed (Participants) | 27 | 35
units on a scale | 0.2 (2.12) | 0.1 (1.97)
Statistical Analysis 1: Comparison: Arm I - Lamotrigine vs Arm II - Placebo; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Brief Pain Inventory (BPI) Average Pain Score [Week 10 Minus Baseline]
Description: The average change in Brief Pain Inventory (BPI) Average Pain scores between baseline and week 10 using Wilcoxon test are reported for each arm below. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: From baseline to week 10
Population: Participants with BPI Average Pain data at both time points available were assessed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Number analyzed (Participants) | 29 | 35
units on a scale | -0.1 (2.15) | -0.8 (2.35)
Statistical Analysis 1: Comparison: Arm I - Lamotrigine vs Arm II - Placebo; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Brief Pain Inventory (BPI) Pain Now Score [Week 10 Minus Baseline]
Description: The average change in Brief Pain Inventory (BPI) Pain Now scores between baseline and week 10 using Wilcoxon test are reported for each arm below. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: From baseline to week 10
Population: Participants with BPI Pain Now data at both time points available were assessed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Number analyzed (Participants) | 30 | 35
units on a scale | -0.1 (2.77) | -0.3 (2.22)
Statistical Analysis 1: Comparison: Arm I - Lamotrigine vs Arm II - Placebo; Test type: Superiority; p = 0.33, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in Brief Pain Inventory (BPI) Pain Relief Score [Week 10 Minus Baseline]
Description: The average change in Brief Pain Inventory (BPI) Pain Relief scores between baseline and week 10 using Wilcoxon test are reported for each arm below. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: From baseline to week 10
Population: Participants with BPI Pain Relief data at both time points available were assessed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Number analyzed (Participants) | 21 | 25
units on a scale | 6.7 (28.34) | 0.4 (30.34)
Statistical Analysis 1: Comparison: Arm I - Lamotrigine vs Arm II - Placebo; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Brief Pain Inventory (BPI) Pain Interference Score [Week 10 Minus Baseline]
Description: The average change in Brief Pain Inventory (BPI) Pain Interference scores between baseline and week 10 using Wilcoxon test are reported for each arm below. The BPI scales range from 0 to 10 with 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Time Frame: From baseline to week 10
Population: Participants with BPI Pain Interference data at both time points available were assessed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Number analyzed (Participants) | 30 | 35
units on a scale | -0.5 (2.17) | -0.8 (2.19)
Statistical Analysis 1: Comparison: Arm I - Lamotrigine vs Arm II - Placebo; Test type: Superiority; p = 0.91, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in POMS Total Score [Week 10 Minus Baseline]
Description: The average change in POMS Total scores between baseline and week 10 using Wilcoxon test are reported for each arm below. The POMS scales are calculated from patient responses on 30 questions asking how they have been feeling during the past week. The scores are all transformed so that 0 is the worst possible value and 100 is the best possible value.
Time Frame: From baseline to week 10
Population: Participants with POMS scales data at both time points available were assessed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
Number analyzed (Participants) | 27 | 34
units on a scale | 1.4 (10.67) | 1.3 (9.09)
Statistical Analysis 1: Comparison: Arm I - Lamotrigine vs Arm II - Placebo; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 10 weeks of the study.
Description: Each CTCAE term is a unique representation of a specific event used for medical documentation/scientific analysis and is a single MedDRA Lowest Level Term (LLT). All AEs are reported below for patients who reported AEs for cycle >0 and grade >0.Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, and appear in the SAE table.
Arm/Group | Arm I - Lamotrigine | Arm II - Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/63
Other Adverse Events (participants affected / at risk) | 26/61 | 24/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Lamotrigine (N=61) | Arm II - Placebo (N=63)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 3 (4)
General symptom (General disorders) | 1 (3) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Pain due to radiation (General disorders) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 14 (54) | 8 (24)
Depressed level of consciousness (Nervous system disorders) | 3 (3) | 2 (3)
Dizziness (Nervous system disorders) | 6 (11) | 11 (30)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (5)
Nystagmus (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 10 (11) | 5 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes